CLINICAL TRIAL: NCT00092885
Title: A Multicenter, Double-Blind, Randomized Study Investigating the Clinical Effect of Montelukast on Allergic Rhinitis in Patients With Seasonal Allergic Rhinitis and Chronic Asthma
Brief Title: An Approved Drug to Study a New Indication for Seasonal Allergic Rhinitis in Patients With Asthma (0476-269)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-269; 2004_025
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Asthma, Bronchial
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0476, montelukast sodium
Drug: Comparator: placebo

SUMMARY:
The purpose of this study is to determine the effect of an approved medication on the symptoms of seasonal allergic rhinitis (a seasonal variety of inflammation of the mucous membrane of the nose) in patients who are experiencing symptoms of seasonal allergic rhinitis and asthma.

DETAILED DESCRIPTION:
The duration of treatment is 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* A 2-year documented history of seasonal allergic rhinitis
* A 1-year documented history of chronic asthma
* Positive allergy testing

Exclusion Criteria:

* Medical history of a lung disorder (other than asthma) or a recent upper respiratory tract infection.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2003-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Daily Rhinitis Symptoms score; the Daytime Nasal Symptoms score and Nighttime Symptoms score

SECONDARY OUTCOMES:
(1) Rhinoconjunctivitis Quality-of-Life Questionnaire overall score; (2) Global Evaluation of Allergic Rhinitis by Patient; (3) Global Evaluation of Allergic Rhinitis by Physician

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Philip G, Nayak AS, Berger WE, Leynadier F, Vrijens F, Dass SB, Reiss TF. The effect of montelukast on rhinitis symptoms in patients with asthma and seasonal allergic rhinitis. Curr Med Res Opin. 2004 Oct;20(10):1549-58. doi: 10.1185/030079904x3348. PMID 15462688